CLINICAL TRIAL: NCT07159750
Title: Real-world Prospective Study on the Use of Anti-CGRP Drugs in Migraine
Acronym: EUREkA
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EOM(AG)008/2024(6234)
Record Dates: First submitted 2025-08-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Episodic Migraine; Chronic Migraine, Headache
Keywords: Migraine; Prevention; Chronic Migraine; Episodic Migraine; galcanezumab; erenumab; fremanezumab; eptinezumab; rimegepant; atogepant
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Calcitonin Gene-Related Peptide Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Migraine Patients: Migraine patients who initiate a CGRP-targeted treatment
  Interventions: Drug: CGRP antibody or gepant

INTERVENTIONS:
Drug: CGRP antibody or gepant — Patients will start anti-CGRP or its receptor antibody or gepants

SUMMARY:
The goal of this observational study is to evaluate clinical differences in patients who received preventive treatment with medication targeting calcitonin gene-related peptide (CGRP) or its receptor: monoclonal antibodies (erenumab, galcanezumab, fremanezumab, eptinezumab) or gepants (rimegepant, atogepant) during a 2-year period observation phase.

DETAILED DESCRIPTION:
It is a 2-year, multicenter observational study. Patients who meet reimbursement criteria according to local regulations and willing to participate in the study will be included. Monoclonal antibodies (erenumab, galcanezumab, fremanezumab, eptinezumab) or gepants (rimegepant, atogepant) will be started and baseline assessment will be conducted. There will be visits every 6 months to assess effectiveness, side-effects, PROMs, and elegibility to continue with the study drug. The observation of patients will last 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Migraine diagnosis according to ICHD-III.
* Prescription of erenumab, galcanezumab, fremanezumab, eptinezumab, atogepant or rimegepant according to prescriptor criteria and reimbursement criteria according to local regulations.
* Signature of informed consent.

Exclusion Criteria:

* Presence of headache different from migraine.
* Active severe psychiatric condition or cognitive impairment which may affect the ability to consent patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Episodic and chronic migraine patients.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Monthly Headache Days and Monthly Migraine Days | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
HIT-6 | Through study completion, an average of 2 years
  Change in HIT-6 (Headache Impact Test) scale, to assess migraine impact.
MIDAS | Through study completion, an average of 2 years
  Change in MIDAS (Migraine Disability Assessment Scale) scale, to assess disability attributed to migraine.
PGIC | Through study completion, an average of 2 years.
  PGIC (Patien Global Impression of Change) scale will be used to assess impression of change in migraine patients.
BAI | Through study completion, an average of 2 years.
  Change in BAI (Beck Anxiety Inventory) scale, to assess anxiety in migraine patients.
BDI-II | Through study completion, an average of 2 years.
  Change in BDI-II (Beck's Depression Inventory, 2nd version) scale, to assess depression in migraine patients.
MSQ Version 2.1 | Through study completion, an average of 2 years.
  Changes in MSQ (Migraine-Specific Quality-of-Life) Version 2.1 scale, to assess patient's quality of life.
WPAI | Through study completion, an average of 2 years.
  Changes in WPAI (Work Productivity and Activity Impairment) questionnaire, to assess how migraine impacts in work and productivity in migraine patients.
ISI | Through study completion, an average of 2 years.
  Changes in ISI (Insomnia Severity Index) scale to assess insomnia in migraine patients.
ASC-12 | Through study completion, an average of 2 years.
  Changes in ASC-12 (Allodynia Symptom Checklist) scale, to assess allodynia in migraine patients.
m-TOQ | Through study completion, an average of 2 years.
  m-TOQ (Migraine Treatment Optimization Questionnaire) scale will be used to assess the effectiveness of migraine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pozo-Rosich, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (26):
- University of Miami, Miller School of Medicine, Miami, Florida, United States
- FLENI, Buenos Aires, Argentina
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Neuromedica, Medellín, Colombia
- Special Hospital for Orthopedics and Rehabilitation "Martin Horvat" Rovinj-Rovigno, Rovinj, Croatia
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - LMU University Hospital, München
- Italy (4):
  - University of L'Aquila, L’Aquila
  - University of Modena and Reggio Emilia, Modena
  - National Neurological Institute C. Mondino Foundation, Pavia
  - IRCCS San Raffaele, Roma
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia
- Neuroclinic Norway, Lillestrøm, Norway
- Wrocław Medical University, Wroclaw, Poland
- Hospital Santa Maria Lisbon, Lisbon, Portugal
- Spain (10):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Fundació Sanitària Mollet, Mollet del Vallès, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital General Universitario de Albacete, Albacete
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - La Paz University Hospital, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No